

#### CONSENTIMIENTO INFORMADO PARA PARTICIPAR EN UN ENSAYO MEDICO

Titulo Simple del HB-adMSC's para Lesiones Neurologicas

Estudio:

Un Ensayo Clínico para Determinar la Seguridad y Eficacia de la Titulo Completo del Terapia de Células Madre Mesenquimales Autólogas de Hope Estudio:

Biosciences para el Tratamiento de Lesiones Cerebrales

Traumáticas y / o Encefalopatía Hipoxica-Isquémica

Patrocinador del

Hope Biosciences Estudio:

Dr. Charles S. Cox, Jr, Profesor, Departamento de Cirugia Pediatrica **Investigator Principal:** 

UTHealth McGovern Medical School

Steven Kosmach, MSN, RN, CCRC, Clinical Trial Program Manager Contacto de Estudio:

713-500-7329

El propósito de este estudio de investigación es probar la seguridad y el beneficio de las infusiones autólogas de células madre mesenquimales derivadas de adiposo, (aquí después denominadas HB-adMSC) como tratamiento para individuos con lesiones cerebrales. "Autólogo" se refiere a las células o teiidos de un individuo, o que provienen de sí mismo. "Adiposo" se refiere a las células de grasa.

Si acepta participar en el estudio, tendrá 7 visitas a la clínica durante un período de 14 meses con cada visita que dura de 2 a 6 horas. También lo contactaremos por teléfono 2 años después de su última infusión de células madre para una breve evaluación de su salud. Habrá una visita adicional para el tejido adiposo (células grasas) que se tomará de una pequeña incisión en el estómago y se procesará a HB-adMSC. Recibirá 3 infusiones de HB-adMSC durante un período de 6 semanas con 14 días que separan las visitas a la infusión. Evaluaremos la seguridad y el beneficio de las infusiones celulares en las visitas de estudio posteriores a la infusión de 6 y 12 meses y en la llamada telefónica de seguimiento de 2 años. Las visitas de estudio se llevarán a cabo en el Hospital de Memorial Hermann Hospital-Texas Medical Center (MHH-TMC) y el hospital de Houston Methodist Research Institute (HMRI). La extracción de células de grasa se realizará en una clínica médica local asociada con Hope Biosciences.

Los riesgos al participar en este estudio incluyen dolor y cicatrices de la incisión abdominal, posible infección, dolor y moretón en el lugar donde se tomaron las muestras de sangre. Los riesgos remotos (extremadamente improbables) incluyen daño a los órganos por la infusión celular y hasta la muerte. Usted no puede beneficiarse directamente al participar en el estudio. El conocimiento obtenido de este estudio puede ayudar a los médicos a desarrollar mejores tratamientos para las personas con lesiones cerebrales.

Su participación es voluntaria; la única alternativa es no participar en este estudio de investigación y continuar con las terapias estándar.

Usted puede optar por no participar en este estudio de investigación o puede optar por dejar el estudio de investigación en cualquier momento. Su decisión no afectará la atención clínica que recibe en la University of Texas Health Science Center en Houston (UTHealth) o Memorial Hermann Healthcare System.

Si usted está interesado en conocer más acerca del estudio clínico, por favor continúe leyendo a continuación.

Nombre de Contacto: Steven Kosmach

713-500-7329 Teléfono:



Está invitado a participar en el protocolo titulado "Un ensayo clínico para determinar la seguridad y eficacia de la terapia de células madre mesenquimales autólogas de Hope Biosciences para el tratamiento de lesiones cerebrales traumáticas y encefalopatía hipoxica-isquémica". Este formulario de consentimiento tiene información importante sobre este estudio para ayudarle a decidir si participa o no en este estudio. Su decisión de participar es voluntaria. Usted puede negarse a participar u optar por dejar de participar, en cualquier momento. La decisión de no participar o dejar de ser parte del proyecto de investigación no cambiará los servicios disponibles para usted en la University of Texas Health Science Center en Houston (UTHealth) y Memorial Hermann Healthcare System.

### ¿Cuál es el propósito de este estudio de investigación?

El propósito de este estudio es investigar la seguridad y el beneficio de HB-adMSC como tratamiento para lesiones neurológicas sub-agudas o crónicas. Hb-adMSC es un producto biológico en investigación y no está aprobado por la Administración de Alimentos y Medicamentos (FDA, por sus siglas en Ingles) aprobado como tratamiento para lesiones neurológicas. Hope Biosciences está pagandole a UTHealth por el trabajo en el estudio.

#### ¿A Quién se le pide que participe en este estudio?

Se le está invitando a participar en el estudio porque usted ha sido diagnosticado con una lesión neurológica sub-aguda o crónica que es poco probable que mejore con el enfoque de atención estándar actual. El estudio se está llevando a cabo en UTHealth e inscribirá a 24 personas.

Una descripción de este ensayo clínico estará disponible en el sitio de internet http://www.clinicaltrials.gov, según lo requiere la Ley de los Estados Unidos. Este no incluirá información que pueda identificarlo. Una vez finalizado el estudio, el sitio de internet incluirá un resumen de los resultados. Puede buscar en este sitio de internet en cualquier momento.

### ¿Que pasara si acepto participar en este estudio? Llamada de Pre-evaluación:

Nuestros procedimientos de selección comienzan con una llamada telefónica para proporcionarle una visión general del estudio y discutir los requisitos de elegibilidad. Está recibiendo este documento de consentimiento informado porque ya ha hablado con el coordinador del estudio y, después de discutir el estudio, ha expresado interés en continuar con los procedimientos de selección. Si, después de revisar este consentimiento, usted todavía está interesado en participar en el estudio, usted o su representante legal (LAR) tendrá que firmar y devolver el consentimiento por correo electrónico o en el sobre prepagado proporcionado. La autorización para la divulgación de información de salud nos permitirá solicitar registros médicos relacionados con su lesión neurológica y determinar su elegibilidad para participar en el estudio.

Programaremos una conferencia telefónica con usted para revisar su historial médico y el consentimiento del estudio para garantizar que todas sus preguntas hayan sido contestadas y usted entienda y acepte las visitas y los procedimientos. La visita de base de referencia se programará en un momento conveniente para usted. Se le proporcionará información sobre las ubicaciones de la clínica y las opciones de estacionamiento para cada visita.

#### Visita 1: Selección

La primera visita de estudio se llevará a cabo en la Unidad de Investigación Clínica (CRU) en MHH y se espera que tome alrededor de 4 horas para completarse. La visita comenzará con



una revisión de este documento de consentimiento para asegurarse que todas sus preguntas han sido contestadas y para verificar su disposición en continuar con el estudio.

#### Usted se someterá a las siguientes evaluaciones/procedimientos:

- Revisión de cualquier cambio en su salud durante el intervalo desde la llamada de conferencia.
- Examen físico y neurológico.
- Se le preguntará sobre su historia clínica, su historia clínica familiar, cualquier medicamento sin receta o recetado tomado en los últimos 30 días, e información demográfica como raza, etnia, empleo y estado civil.
- Signos vitales que incluyen presión arterial, frecuencia cardíaca, temperatura, frecuencia respiratoria y saturación de oxígeno.
- Recolección de muestras de sangre (aproximadamente 4 cucharadas) para pruebas clínicas de laboratorio de rutina que miden su salud general (CBC con paneles de diff, metabólicos, coagulación y función renal), prueba de laboratorio de investigación, y prueba de embarazo para mujeres en edad fértil.
- Radiografia del tórax.
- Exámenes y evaluaciones estandarizadas para medir su grado de discapacidad por la lesión cerebral.

El equipo de investigación revisará los resultados de las pruebas de los procedimientos mencionados anteriormente. Si los resultados son anormales de la prueba, como una radiografía de tórax que sugiere que hay una infección respiratoria puede requerir que la visita se cancele y se reprograme para después. Siempre existe el potencial de que la nueva información de los resultados de la prueba podría impedir su participación en el estudio. Un coordinador del estudio lo llamará dentro de las 24 horas de la visita para programar los próximos procedimientos de estudio o discutir los resultados de la prueba impidiendo su participación continua en el estudio.

Si usted es elegible para continuar en el estudio, programaremos la visita de extracción de células de grasa con Hope Biosciences. En la visita, se utilizará un anestésico local para adormecer la piel del abdomen, el flanco o la zona de la cadera. Luego se hará una pequeña incisión para colectar alrededor de 2 cucharadas de tejido adiposo, y luego se cerrará y cubrirá con una gasa estéril. Se le vigilará de cerca durante el procedimiento corto. El coordinador del estudio se pondrá en contacto con usted al día siguiente de la extracción de grasa para evaluar su recuperación.

Hope Biosciences procesará sus células de grasa en HB-adMSC durante un período de 5 a 7 semanas. Existe la posibilidad remota de que la infusión de HB-adMSC no cumpla con los estrictos criterios de liberación de Hope Biosciences. Las razones incluyen una cantidad insuficiente de células madre para entregar la dosis del objetivo o la contaminación del producto. Si ocurre un evento improbable como este, se le contactará inmediatamente y se le dará la opción de repetir la visita de extracción de grasa o retirarse del estudio.

### Visita 2: Imagen de Referencia

La visita para la imagen(es) de referencia se llevará a cabo en el HMRI y se programará dentro de los 10 días posteriores a su visita de selección. Se espera que la visita tome unas 5 horas en completarse.



Fecha de Versión de Documento: 7 SEP 2021

#### Usted se someterá a las siguientes evaluaciones/procedimientos:

- Revisión de cualquier cambio de intervalo en su salud desde la última visita.
- Examen físico y neurológico.
- Signos vitales que incluyen presión arterial, frecuencia cardíaca, temperatura, frecuencia respiratoria y saturación de oxígeno.
- Se repetirá una prueba de embarazo para mujeres en edad fértil.
- Inserción de una aguja intravenosa (IV) en una vena de la mano o del antebrazo.
- Una tomografía por emisión de positrones (PET)/Imagen por Resonancia Magnética (MRI, por sus siglas en Ingles).
- Instrucciones sobre la administración de Lovenox por invección durante 7 días a partir del día antes de cada visita a la infusión y completar el registro de medicamento de Lovenox.

Una tomografía por emisión de positrones (PET) es una técnica de imagen que utiliza un radio marcador diseñado para unirse o "pegarse" a tipos específicos de células en el cuerpo humano. Los radio marcadores contienen una cantidad muy pequeña de radioactividad y se administran mediante una inyección intravenosa inmediatamente antes de la tomografía por emisión de positrones. La imagen PET a continuación mide la ubicación y la cantidad de radio marcador. [11C] ER-176 es un radio marcador diseñado para unirse a un tipo de células cerebrales llamadas microglía. Las células de microglía desempeñan un papel importante en la sanación cerebral después de una lesión.

La imagen por resonancia magnética (IRM) utiliza un gran imán y ondas de radiofrecuencia para crear imágenes de estructuras internas del cuerpo; por lo que no hay exposición a la radiación.

Para ambos escaneos, se le colocará sobre una mesa acolchada y se le pedirá que se acueste boca arriba. Usted podrá comunicarse con el personal de imágenes durante las exploraciones y ellos podrán verlo y escucharlo. En varios puntos de tiempo se le pedirá que se quede perfectamente quieto mientras la máquina está escaneando. El personal de radiología contacta rutinariamente a los pacientes las 24 horas después de los exámenes por imágenes para una breve evaluación de la salud del paciente.

#### Visitas 3 a 5: Infusiones HB-adMSC

Tendrá tres visitas para la infusión durante un período de 6 semanas con 14 días (+/- 2 días) separando las infusiones. Cada visita se llevará a cabo en la CRU en MHH y tardará alrededor de 6 horas en completarse. Recibirá una llamada de recordatorio del equipo de estudio para comenzar las invecciones de Lovenox el día antes de la visita.

#### Usted se someterá a las siguientes evaluaciones/procedimientos:

- Revisión de cualquier cambio en su salud durante el intervalo desde la última visita de estudio,
- Revisión del registro de medicamentos de Lovenox,
- Signos vitales que incluyen presión arterial, frecuencia cardíaca, temperatura, frecuencia respiratoria y saturación de oxígeno.
- Recolección de muestras de sangre (aproximadamente 2 cucharadas) para laboratorios clínicos de rutina que evalúan su salud general (CBC con paneles de diff, metabólicos, coagulación y función renal), y prueba de embarazo para mujeres en edad fértil.
- Se insertará una aquia intravenosa en una vena de la mano o del antebrazo para la infusión de las HB-adMSC autólogos.

Nombre de Contacto: Steven Kosmach 713-500-7329 Teléfono:



Fecha de Versión de Documento: 7 SEP 2021

Supervisaremos sus signos vitales de cerca durante la infusión y durante las próximas 4 horas después de la infusión. El equipo de investigación se pondrá en contacto con usted por teléfono al día siguiente de la infusión para una breve evaluación de su salud desde que salió del hospital.

#### Visita 6: Seis Meses después de la Infusión:

Se le pedirá que regrese seis meses después de la última infusión HB-adMSC. La visita se llevará a cabo en ambos lugares el CRU y el HMRI y se espera que tome acerca de 8 horas para completar. La visita puede programarse para un periodo de dos días.

### <u>Usted se someterá a las siguientes evaluaciones/procedimientos:</u>

- Revisión de cualquier cambio en su salud durante el intervalo desde la última visita de estudio,
- Examen fisico y neurologico,
- Signos vitales que incluyen presión arterial, frecuencia cardíaca, temperatura, frecuencia respiratoria y saturación de oxígeno.
- Recolección de muestras de sangre (aproximadamente 2 cucharadas) para laboratorios clínicos de rutina que evalúan su salud general (CBC con paneles de diff, metabólicos, coagulación y función renal), y prueba de embarazo para mujeres en edad fértil.
- Recolección de muestras de sangre (aproximadamente 1 cucharada) para pruebas de laboratorio de investigación.
- Un escan del cerebro de PET/MRI.
- Exámenes y evaluaciones estandarizados para medir su grado de discapacidad de la lesión cerebral.

#### Visita 7: Un Año después de la Infusión

La visita del estudio se llevará acabo en el CRU y se espera que tome acerca de 2 horas para completar.

#### Usted se someterá a las siguientes evaluaciones/procedimientos:

- Revisión de cualquier cambio en su salud durante el intervalo desde la última visita de estudio,
- Examen fisico y neurológico,
- Signos vitales que incluyen presión arterial, frecuencia cardíaca, temperatura, frecuencia respiratoria y saturación de oxígeno.
- Recolección de muestras de sangre (aproximadamente 2 cucharadas) para laboratorios clínicos de rutina que evalúan su salud general (CBC con paneles de diff, metabólicos, coagulación y función renal), y prueba de embarazo para mujeres en edad fértil.
- Recolección de muestras de sangre (aproximadamente 1 cucharada) para pruebas de laboratorio de investigación.
- Radiografia del tórax.
- Exámenes y evaluaciones estandarizados para medir su grado de discapacidad de la lesión cerebral.

### Llamada Telefónica de Seguimiento Dos Años Después

Un miembro del equipo de investigación se pondrá en contacto con usted por teléfono 2 años después de su última infusión de células madre para determinar si ha tenido algún problema de



Fecha de Versión de Documento: 7 SEP 2021

salud desde su última visita de estudio. La llamada telefónica será breve y no tardará más de 10 minutos en completarse.

# ¿Cuánto tiempo va a estar usted en el estudio?

Si acepta participar en este estudio, su participación durará unos 14 meses y consta de 7 visitas de estudio en el MHH y/o el HMRI y 1 visita en una clínica asociada con Hope Biosciences.

#### ¿Qué opciones tiene usted aparte de este estudio?

Usted puede continuar con terapias convencionales y/o identificar otros ensayos clínicos para los cuales usted puede ser elegible.

### ¿Cuáles son los riesgos al tomar parte en este estudio?

#### Extracción de Muestras de Sangre:

La obtención de muestras de sangre puede causar molestias menores, sensación de mareo, desmayo, moretones, coagulación y sangrado del sitio del pinchazo de la aguja y, en raras ocasiones, infección.

#### Extracción de Grasa e Infusiones HB-adMSC:

El procedimiento para recolectar grasa del estómago dejará una pequeña cicatriz, y usted puede experimentar molestias por el procedimiento quirúrgico. El área alrededor de la incisión se adormecerá con anestesia local para minimizar las molestias y el procedimiento se realizará utilizando una técnica estéril para minimizar el riesgo de infección. Debido a que la infusión de células madre es un producto de su cuerpo, no esperamos ninguna reacción mala que a veces puede ocurrir cuando se obtienen células madre de otro individuo. Para minimizar cualquier posible reacción, se le administrarán dos medicamentos (Benadryl y Solumedrol) antes de la infusión. Ambos medicamentos están aprobados por la (FDA, por sus siglas en Ingles). Los riesgos potenciales de la infusión intravenosa de HB-adMSC's incluyen coágulos sanguíneos, infección, dificultad respiratoria/insuficiencia, lesión hepática, lesión neurológica, crecimiento tumoral, insuficiencia orgánica y hasta la muerte.

#### Lovenox:

Para minimizar el riesgo potencial de coágulos sanguíneos, se le administrara Lovenox. Los riesgos potenciales de Lovenox incluye irritación, dolor, moretones, enrojecimiento o hinchazón en el sitio de la invección.

### Imagen de PET:

Durante la exploración recibirá la cantidad de radioactividad similar a la que ha estado expuesto en los últimos 15 meses de fuentes de fondo naturales. Se estima que los niveles seguros de exposición a la radiación para los seres humanos son de aproximadamente 50 milisieverts (mSv) en el transcurso de 1 año. La exposición a la radiación por imagen de PET es de aproximadamente 20 mSv para ambos escaneos y esto está dentro del límite de seguridad.

#### Imagen por Resonancia Magnética (IRM):

No se requiere radiación ni medios de contraste para la resonancia magnética cerebral. Algunas personas encuentran incómodo el espacio estrecho del escáner. Los medicamentos están disponibles para personas con claustrofobia. Las máquinas de resonancia magnética hacen ruidos fuertes de golpes y clics durante los escaneos. Los auriculares estarán disponibles para su comodidad. Los imanes grandes utilizados para la imagen de RM pueden interactuar con objetos metálicos como aparatos dentales o dispositivos implantados. Se le evaluara cuidadosamente para la presencia de objetos metálicos en o en su cuerpo antes de la IRM.

Nombre de Contacto: Steven Kosmach Teléfono: 713-500-7329

Fecha de Versión de Documento: 7 SEP 2021

Es posible que nos enfrentemos con problemas inesperados e imprevistos relacionados con la infusión de HB-adMSC.

Vacunaciones de Covid-19 Durante la Participación en el Estudio Clínico

Recomendamos altamente a los sujetos que reciban las vacunas para el Covid-19. Sin embargo, se sabe que las vacunas en general causan una respuesta inflamatoria temporal que puede alterar los resultados de las pruebas del estudio y las infusiones de células madre. Le pediremos que no le administren una vacuna para el Covid-19 o una inyección de refuerzo dos semanas antes de las visitas de imágenes cerebrales y dos semanas antes y después de la visita de infusión de células madre.

#### Embarazo/ Control de Natalidad:

Los efectos de HB-adMCS's en los órganos reproductores humanos y los bebés por nacer no se han estudiado y pueden ser perjudiciales de maneras que actualmente no conocemos.

**Para Mujeres:** Si usted está embarazada, planeando quedar embarazada, o está amamantando a un bebe, usted no puede participar en este estudio.

### Para Mujeres & Hombres:

Debe utilizar al menos un método anticonceptivo altamente eficaz durante el estudio. Si ya está usando anticonceptivos, el equipo de investigación le informará si su método anticonceptivo actual es aceptable durante el estudio. Los métodos anticonceptivos aceptables incluyen los siguientes métodos altamente efectivos:

- Anticonceptivos hormonales.
- Dispositivo intrauterino (DIU).
- Esterilización quirúrgica (atadura u obstrucción de las trompas de Falopio, vasectomía).
- Abstinencia sexual verdadera (no tener relaciones sexuales heterosexuales durante el estudio si esto está en conformidad con su estilo de vida preferido y habitual).

Usted debe notificar al equipo de estudio inmediatamente si usted, o para los hombres, su pareja queda embarazada durante el estudio.

## ¿Cuáles son los beneficios al participar en este estudio?

Usted no podrá beneficiarse directamente al participar en el estudio. El conocimiento obtenido de este estudio puede ayudar a los médicos a desarrollar mejores tratamientos para las personas con lesiones cerebrales.

# ¿Puedo dejar de tomar parte en este estudio?

Usted puede decidir dejar de participar en el estudio en cualquier momento. Para retirarse del estudio, póngase en contacto con el Dr. Cox llamando al teléfono 713-500-7300.

Su médico o Hope Biosciences pueden interrumpir el estudio en cualquier momento. Su médico puede detener su participación en el estudio si su condición empeora, o si usted no cumple con todos los requisitos del estudio, y/o el estudio no es lo mejor para de usted. Si se interrumpe su participación en el estudio, su médico analizará otras opciones para su tratamiento.

Si deja de participar en este estudio, la información ya recopilada sobre usted seguirá utilizándose en el análisis de datos. Sin embargo, no se recopilará más información sin su permiso.

Durante su participación en este estudio, el equipo de estudio le notificará de nueva información que puede estar disponible y podría afectar su disposición en permanecer en el estudio.



Fecha de Versión de Documento: 7 SEP 2021

## ¿Qué sucede si usted resulta lesionado durante el estudio?

Si necesita tratamiento médico para una enfermedad o lesión que es el resultado directo de tomar el producto de estudio, Hope Biosciences pagará los costos razonables y rutinarios de dichos tratamientos si se cumplen las siguientes condiciones:

- La enfermedad o lesión fue el resultado de la participación en el estudio.
- El costo del tratamiento o cualquier parte de los costos no está cubierto por ningún otro seguro de salud, programa de salud del gobierno u otros que proporcionen cobertura para atención médica.

No hay pago ni reembolso disponible por cosas tales como condiciones preexistentes, enfermedades o enfermedades totalmente ajenas al estudio, salarios perdidos, daños a la propiedad, discapacidad o malestar. Usted o su compañía de seguros serán responsables del pago de cualquier prueba o cuidado realizado fuera del alcance del estudio.

Si usted sufre alguna lesión como resultado de participar en este estudio de investigación el patrocinador de este estudio, Hope Biosciences, pagará los gastos médicos razonables y necesarios si la lesión es un resultado directo de tomar el medicamento de estudio o someterse a unos procedimientos de estudio, y que no sea debido al curso natural de cualquier enfermedad subvacente o proceso de tratamiento.

Usted debe reportar cualquier lesión de este tipo al Dr. Cox al teléfono 713-500-7300 y al Comité para la Protección de los Sujetos Humanos al teléfono 713-500-7943. Usted no renunciará a ninguno de sus derechos legales mediante la firma de este formulario de consentimiento.

Si usted es tratado por una lesión de investigación pagada por Hope Biosciences, Hope Biosciences o su representante recopilará su nombre, fecha de nacimiento, género y número de reclamo de seguro médico de Medicare o número de seguro social para determinar su estado de Medicare. Si usted es beneficiario de Medicare, Hope Biosciences reportará el pago y la información sobre el estudio en el que se encuentra a los Centros de Servicios de Medicare y Medicaid, de acuerdo con los requisitos de informes de (CMS, por sus siglas en Ingles). Hope Biosciences no utilizará esta información para ningún otro propósito.

### ¿Cuáles son los costos asociados al participar en este estudio?

El patrocinador del estudio pagara por todas las visitas y procedimientos relacionados con el estudio.

Si usted recibe un cobro que usted cree que está relacionado con tomando parte en este estudio de investigación, por favor contacte al Dr. Cox al teléfono 713-500-7300 o a su coordinador de estudio al teléfono 713-500-7329.

Usted recibirá \$20 por cada visita de estudio para cubrir el costo del estacionamiento.

### ¿Que pasara con mis muestras de mi sangre y tejido graso?

Las muestras de sangre y tejido graso solo se utilizarán para pruebas específicas que sean necesarias para este estudio. Todas las muestras serán destruidas al concluir los exámenes de prueba a menos que usted dé permiso para su uso futuro.

| ☐ Si ☐ | No | Yo doy mi consentimiento para muestras de tejido sobrante que se utilizaran |
|---|---|---|
| | | para investigaciones futuras conducidas por Hope Biosciences. |



#### ¿Podemos contactarlo en el futuro?

| Podemos | contactarlo | en el | futuro | acerca | de | otros | estudios | de | investigación | que | usted | podría |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| estar interes | sado? | | | | | | | | | | | |

## ¿Cómo se protegerán la privacidad y confidencialidad?

Si No Yo doy mi consentimiento para contacto futuro.

Su privacidad es importante y su participación en este estudio se mantendrá confidencial. Sin embargo, no se puede garantizar la confidencialidad absoluta.

Si firma este documento, usted da permiso a UTHealth y Memorial Hermann Healthcare System para usar y divulgar (liberar) su información médica. La información de salud que podemos usar o divulgar para esta investigación incluye toda la información en su expediente médico, los resultados de exámenes físicos, historial clínico y resultados de pruebas de laboratorio y diagnóstico. Por favor, entienda que la información de salud utilizada y divulgada puede incluir información relacionada con la infección por VIH, abuso de drogas, abuso de alcohol, salud conductual y atención psiguiátrica. La información de identificación que divulgamos a Hope Biosciences se limitará en la medida de lo posible según lo exijan las regulaciones y las leyes que rigen las instalaciones de laboratorio de células madre.

Es posible que las leyes federales de privacidad (como la Regla de Privacidad) no exijan a los coordinadores, investigadores y personal administrativo que reciban su información de salud que protejan su información de salud y puedan compartir su información con otras personas sin su permiso, si lo permiten las leyes que los rigen. Usted no será identificado personalmente en ningún informe o publicación que pueda resultar de este estudio. Si toda la información que lo identifica o puede identificarlo se elimina de su información médica, la información restante ya no estará sujeta a esta autorización y podrá ser utilizada o divulgada para otros fines.

Los representantes de las organizaciones enumeradas a continuación verán su nombre y otros identificadores personales cuando revisen sus registros de investigación y expedientes médicos con el fin de verificar los datos del estudio.

- Representantes de UTHealth y/o Memorial Hermann Health System
- Representantes del patrocinador de esta investigación, incluidas las organizaciones de investigación por contrato y el Monitor de Seguridad Medica
- Miembros de la Junta de Monitoreo de Datos y Seguridad (un grupo independiente de expertos que revisa los datos de este estudio para asegurarse de que los participantes estén seguros y que los datos de investigación sean fiables)
- Representantes de la Administración de Alimentos y Fármacos de los Estados Unidos (FDA, por sus siglas en Ingles)

Tenga en cuenta que no tiene que firmar esta Autorización, pero si no lo hace, no puede participar en este estudio de investigación. UTHealth y Memorial Hermann Health System no pueden denegar el tratamiento o negarse a tratarlo si no firma esta Autorización.

Puede cambiar de opinión y revocar (recuperar) esta Autorización en cualquier momento. Incluso si revoca esta Autorización, los investigadores todavía pueden usar o divulgar información de salud que ya han obtenido sobre usted según sea necesario para mantener la integridad o fiabilidad de la investigación actual. Para revocar esta Autorización, debe comunicarse con el Dr. Cox por escrito a: UTHealth, 6431 Fannin Street, MSB 5.324, Houston, TX 77030.

Esta Autorización expirará 15 años después de finalizar el estudio.

Nombre de Contacto: Steven Kosmach 713-500-7329 Teléfono:



### ¿Con quién puedo ponerme en contacto si tengo preguntas sobre el estudio?

Si tiene preguntas en cualquier momento sobre este estudio de investigación, no dude en ponerse en contacto con el Dr. Cox al teléfono 713-500-7300, ya que estará encantado de responder a sus preguntas. Puede ponerse en contacto con el equipo de estudio para discutir problemas, reportar lesiones, expresar sus preocupaciones, obtener información además de hacer preguntas sobre la investigación.

El Comité para la Protección de los Sujetos Humanos del Centro de la University of Texas Health Science ha revisado este estudio de investigación. Puede ponerse en contacto con ellos para cualquier pregunta sobre sus derechos como sujeto de investigación, y para discutir cualquier inquietud, comentario o queja sobre participar en un estudio de investigación al teléfono (713) 500-7943.

#### **FIRMAS**

Firme a continuación sólo si entiende la información que se le ha dado sobre la investigación y elige participar en este estudio de investigación. Asegúrese de que todas sus preguntas han sido respondidas. Si decide participar en este estudio de investigación, se le dará una copia de este formulario de consentimiento firmado.

| Nombre Impreso del Participante | Firma del Participante | Fecha | Hora |
|---|---|---|---|
| Nombre Impreso del<br>Representante Legal | Firma del Representante Legal | Fecha | Hora |
| Nombre Impreso de la persona que obtiene el consentimiento | Firma de la persona que obtiene el Consentimiento | Fecha | Hora |

Nombre de Contacto: Steven Kosmach Teléfono: 713-500-7329 IRB NUMBER: HSC-MS-19-0685
UTHealth
The University of Ten Houston
The University of Ten Houston